CLINICAL TRIAL: NCT03472274
Title: The DUTRENEO Trial: A Prospective Study to Individualize the Approach With DUrvalumab (MEDI4736) and TREmelimumab in NEOadjuvant Bladder Cancer Patients.
Brief Title: Durvalumab (MEDI4736) and TREmelimumab in NEOadjuvant Bladder Cancer Patients (DUTRENEO)
Acronym: DUTRENEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion CRIS de Investigación para Vencer el Cáncer (Other)
Collaborators: AstraZeneca (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DUTRENEO; 2017-002246-68 (EudraCT Number)
Record Dates: First submitted 2018-03-14; First posted 2018-03-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — durvalumab; tremelimumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cisplatin-based neoadjuvant chemotherapy (Active Comparator): Patients allocated to the control arm will receive any of the following cisplatin based neoadjuvant treatment:
  Regimen 1: Gemcitabine + Cisplatin Regimen 2: Methotrexate + Vinblastine + Doxorubicin + Cisplatin Regimen 3: Gemcitabine + Paclitaxel + Cisplatin
  Interventions: Drug: Cisplatin-based neoadjuvant chemotherapy
- Durvalumab plus Tremelimumab (Experimental): Patients randomized to experimental arma will receive 28-day treatment cycle x 3 cycles of Durvalumab + Tremelimumab 75 mg every 4 weeks
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab 1500 mg every 4 weeks x 3 cycles
  Arms: Durvalumab plus Tremelimumab
Drug: Tremelimumab — Tremelimumab 75 mg every 4 weeks x 3 cycles
  Arms: Durvalumab plus Tremelimumab
Drug: Cisplatin-based neoadjuvant chemotherapy — Regimen 1: 21-day treatment cycle x 3 cycles.
  * Gemcitabine 1,000-1,200 mg/m2 intravenously on days 1 and 8 every 21 days.
  * Cisplatin 70 mg/m2 intravenously on day 1 every 21 days. Regimen 2: ddMVAC 14-day treatment cycle x 4 doses.
  * Methotrexate 30mg/m2 intravenously on day 1
  * Vinblastine 3mg/m2 intravenously on day 2
  * Doxorubicin 30mg/m2 intravenously on day 2
  * Cisplatin 70mg/m2 intravenously on day 2 Granulocyte colony-stimulating factor (G-CSF) for 7 consecutive days (days 4 through 10).
  Regimen 3: 21-day treatment cycle x 3 cycle
  * Gemcitabine 1,000 mg/m2 intravenously on day 1 and 8
  * Paclitaxel 80 mg/m2 intravenously on day 1 and 8
  * Cisplatin 70mg/m2 intravenously on day 1
  Other Names: Standard of care (SoC)
  Arms: Cisplatin-based neoadjuvant chemotherapy

SUMMARY:
In the treatment of localized/locally advanced urothelial cancer, there are several questions that have not yet been resolved, such as the limited benefit of cisplatin-based chemotherapy in the adjuvant or neoadjuvant context, the difficulty in establishing which groups actually benefit from either perioperative treatment and what are the molecular markers that could help us predict the response to this treatment to allow a better selection of patients. On the other hand, not all patients are candidates for cisplatin-based chemotherapy and carboplatin is not comparable in activity, so there is an urgent need to find other drugs that may offer a therapeutic opportunity to these patients.

In the context of metastatic disease, immunotherapy has been able to modify the natural history of this disease, administered as monotherapy, but the combination with double immune checkpoint inhibitors is also being evaluated with promising results. Even this therapeutic strategy is being advanced to the context of adjuvant and neoadjuvant treatment of urothelial tumors. In this sense, on the one hand, the present study, as a research in the neoadjuvant setting, constitutes the opportunity to define molecular phenotypes in bladder cancer since the design of this study will allow both, to evaluate the efficacy of the drug when the tumor is operable and to carry out an extensive analysis of biomarkers in the tumor tissue of these patients with an in-vivo evaluation of immune-based therapy activity. On the other hand, it allows to evaluate a strategy of double-immune checkpoint inhibitors that has already demonstrated activity in metastatic disease and, taking into account, the modest benefit of standard chemotherapy in the perioperative context: platinum-based neoadjuvant chemotherapy in patients with muscle-invasive bladder cancer (MIBC) Modest increase in overall survival, but only a subset of eligible patients are eligible to receive it. In addition, radical cystectomy alone, in MIBC patients, presents a 5-year relapse rate of 10-50%.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects; age ≥ 18 years at the time of study entry.
2. Subjects must provide written informed consent prior to performance of any protocol-related procedures, including screening evaluations and must be willing to comply with treatment and follow up.
3. Subjects must have histologic documentation of transitional cell carcinoma of the urothelium (including the urinary bladder, ureter, urethra and renal pelvis) of the urinary tract (cystoscopy and biopsy or positive cytology).
4. Patients must have confirmed cT2-T4 N0-1 M0 (TNM classification).
5. Archival tumour samples for biomarker research in formalin-fixed and paraffin-embedded blocks.
6. Body weight >30kg
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Life expectancy of at least 12 weeks
9. Adequate organ function as determined by:

   a) Hematological (without growth factor or transfusion support within 28 days prior to first dose of investigational product)
   * Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L).
   * Platelets ≥ 100,000/mm3 (≥ 100 GI/L)
   * Hemoglobin ≥ 9 g/dL (≥ 90 g/L)
10. Hepatic:

    1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN.
    2. Total bilirubin ≤ 1.5 × the upper limit of normal. For subjects with Gilbert's disease ≤ 3 mg/dL (≤ 51.3 μmol/L).
11. Renal:

    a) Calculated CrCl or 24-hour urine CrCl>40 mL/min or Calculated creatinine clearance CL>40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
12. Fasting serum triglycerides ≤ 2.5 × upper limit of normal AND total cholesterol ≤ 300 mg/dL (≤ 7.75 mmol/L). Lipid-lowering medication is allowed.
13. HbA1c ≤ 8%.
14. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.

Exclusion Criteria:

1. Histology of pure adenocarcinoma, pure squamous cell carcinoma, or predominant small cell carcinoma or sarcomatoid features in the tumor sample.
2. Evidence of any metastatic lesion outside the primary tumour site identified in the radiological evaluation.
3. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids or local steroid injections (eg, intra-articular injection).
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent.
   * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
4. Previous therapy with PD-1, PD-L1 or CTLA-4 inhibitors, including durvalumab and tremelimumab.
5. Any concurrent chemotherapy, immunotherapy (IMT), or biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
6. History of severe allergic reactions (ie, Grade 4 allergy, anaphylactic reaction from which the subject did not recover within 6 hours of institution of supportive care) to any unknown allergens or any components of the study drug formulations.
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
8. Major surgery within 4 weeks of study randomization.
9. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
10. Prior radiation therapy to >25% of the bone marrow.
11. Current treatment on another clinical trial.
12. Diagnosis of any second malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
13. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident including transient ischemic attack, or pulmonary embolus.
14. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 electrocardiograms (ECGs).
15. Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

    * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
    * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
16. Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy)
17. Current treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
18. History of active primary immunodeficiency
19. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), hepatitis B (known positive hepatitis B virus (HBV) surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV Ribonucleic acid (RNA).
20. Known positive for human immunodeficiency virus (HIV), chronic or active hepatitis B or C or active hepatitis A.
21. Receipt of live, attenuated vaccine within 30 days prior to the first dose of investigational products.
22. Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to randomization.
23. Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
24. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
25. History of leptomeningeal carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Antitumor activity | 20 weeks
  Evidence of residual disease based on pathological review of the surgical specimen

SECONDARY OUTCOMES:
Overall Objective Response Rate | 20 weeks
  Number of complete response (CR) or partial response (PR) according to RECIST v1.1.
Disease Free Survival | 2 years
  Number of disease recurrences according to RECIST v1.1 or death due to any cause, whichever occurs first
Overall Survival | 2 years
  Number of deaths due to any cause
Incidence of Adverse Events | 20 weeks
  Number of Adverse Events per patient using the National Cancer Institute Common Toxicity Criteria (CTC)

OTHER OUTCOMES:
Biomarkers of response | 20 weeks
  Candidate biomarkers of response in peripheral blood and tumor biopsy specimens that may prospectively identify subjects most likely to respond to treatment
Biomarker expression | 20 weeks
  Changes in biomarker expression in pre-treatment and post-treatment tumor samples of patients treated.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Grande, MD, Principal Investigator — MD Anderson Cancer Center Madrid
Locations (11):
- Spain (11):
  - ICO Badalona, Badalona
  - Hospital Clinic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - ICO L'Hospitalet, L'Hospitalet de Llobregat
  - Hospital 12 de Octubre, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Marqués de Valdecilla, Santander
  - Instituto Valenciano de Oncología, Valencia

REFERENCES:
- [Derived] Sibai M, Cervilla S, Grases D, Musulen E, Lazcano R, Mo CK, Davalos V, Fortian A, Bernat A, Romeo M, Tokheim C, Barretina J, Lazar AJ, Ding L; DUTRENEO Study Investigators; Grande E, Real FX, Esteller M, Bailey MH, Porta-Pardo E. The spatial landscape of cancer hallmarks reveals patterns of tumor ecological dynamics and drug sensitivity. Cell Rep. 2025 Feb 25;44(2):115229. doi: 10.1016/j.celrep.2024.115229. Epub 2025 Jan 24. PMID 39864059